CLINICAL TRIAL: NCT00004093
Title: A Phase I-II Study of Induction Chemotherapy With Carboplatin and Gemcitabine, Followed by Chemoradiotherapy With Paclitaxel and Vinorelbine for Patients With Locally Advanced Non-Small Cell Lung Cancer
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Stage III Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Original Principal Investigator left the institution.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 99L1; NU-99L1; NCI-G99-1585
Record Dates: First submitted 1999-12-10; First posted 2003-11-04 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Gemcitabine; Paclitaxel; Vinorelbine; Radiotherapy

INTERVENTIONS:
Drug: carboplatin — Carboplatin will be dosed at a target AUC of 5, and will be given on day 1 of each cycle
Drug: Gemcitabine — Gemcitabine will be given at 1000 mg/m2 IV over 30 minutes on days 1 and 8 of each 21-day cycle of induction chemo (following carboplatin on day 1).
Drug: paclitaxel — Paclitaxel will be given on day 1 of each week for 6 weeks at a dose of 50 mg/m2.
Drug: vinorelbine — Vinorelbine will be given on day 1 of each week for 6 weeks at a starting dose of 10 mg/m2, escalating up to 15 mg/m2 if no dose limiting toxicities are observed.
Radiation: radiation therapy — Radiation will be given at a dose ranging between 45 to 66 Gy, depending on patient-specific characteristics.
Drug: Navelbine — Navelbine will be administered at a dose of 10-15 mg/m2 in 100 cc NS to be administered over 10 minutes I.V. (one dose weekly during radiation therapy)
Drug: Taxol — Taxol will be administered at a dose of 50 mg/m2 in 250 cc of NS or D5W over 60 minutes, following Navelbine (one dose weekly during radiation therapy)

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy and radiation therapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy plus radiation therapy in treating patients who have stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility of the concurrent chemoradiotherapy regimen of paclitaxel and vinorelbine with standard chest radiotherapy in patients with locally advanced non-small cell lung cancer. II. Determine the maximum tolerated dose and dose limiting toxicities of this regimen in this patient population. III. Determine the radiologic response rate of induction chemotherapy with carboplatin and gemcitabine in this patient population. IV. Evaluate the pathologic response rate in patients undergoing resection. V. Evaluate the time to progression, overall survival, and quality of life in this patient population.

OUTLINE: This is a dose escalation study of vinorelbine. Patients receive induction chemotherapy consisting of carboplatin IV over 30 minutes on day 1 followed by gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks for 2 courses. At 2 weeks following completion of induction chemotherapy, patients receive vinorelbine IV over 10 minutes followed by paclitaxel IV over 60 minutes weekly and radiotherapy daily for 5 consecutive days a week on weeks 1-6. Following initial induction chemotherapy, patients with stable or regressive disease may receive an additional 2-4 courses of carboplatin and gemcitabine at investigator's discretion. At approximately 2-6 weeks following completion of chemoradiotherapy, patients with resectable/operable disease undergo surgical resection. Cohorts of 3-6 patients receive escalating doses of vinorelbine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 3 of 6 patients experience dose limiting toxicity. Quality of life is assessed in all patients. Patients are followed at 1 month.

PROJECTED ACCRUAL: A total of 38-47 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed stage IIIA or IIIB non-small cell lung cancer Pathologic staging of mediastinal lymph nodes required (N2, N3) Bidimensionally measurable disease by x-ray, CT scan, or MRI OR Evaluable disease (e.g., pulmonary infiltrate evaluable on x-ray) No malignant pleural effusions

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 8 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 3 times ULN Renal: Creatinine no greater than 1.5 times ULN OR Creatinine clearance at least 50 mL/min Cardiovascular: No active cardiac ischemia No congestive heart failure Other: No significant active infection No other severe complicating medical illness (e.g., severe neurologic or psychiatric disease that would prevent compliance) No concurrent malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior pelvic or thoracic radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 1999-08; Primary Completion 2002-02 (Actual); Study Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of the combination therapies | After each cycle of therapy
  Toxicity will be assessed for each patient after each cycle of therapy. The maximum tolerated dose (MTD) will be the dose level prior to the dose in which greater than one-third of patients experience a dose-limiting toxicity.
Determine the radiologic response rate of the combined study therapies | After every 2 cycles of study therapy
  Patients will have a radiographic work-up (in the form of a chest CT) after every 2 cycles of therapy to assess tumor response to the study therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A. Masters, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Argiris A, Liptay M, LaCombe M, Marymont M, Kies MS, Sundaresan S, Masters G. A phase I/II trial of induction chemotherapy with carboplatin and gemcitabine followed by concurrent vinorelbine and paclitaxel with chest radiation in patients with stage III non-small cell lung cancer. Lung Cancer. 2004 Aug;45(2):243-53. doi: 10.1016/j.lungcan.2004.02.008. PMID 15246197